CLINICAL TRIAL: NCT05046522
Title: A Double-blind Randomised Controlled Study to Evaluate the Effectiveness of Orally-dosed Palmitoylethanolamide (PEA) Compared to Placebo for Reducing Pain Severity and Duration of Migraines in Otherwise Healthy Participants Aged 18 Years and Older.
Brief Title: A Study Evaluating the Effectiveness of PEA Compared to Placebo for Reducing Pain Severity and Duration of Migraines.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIGLEV-21
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2022-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palmitoylethanolamide sold as Levagen + (Experimental): Palmitoylethanolamide in capsule form - taken as a 700mg (2 x 350mg) dosage at onset of migraine and if unresolved at 2 hours post onset a second dose of 700mg (2 x 350mg)
  Interventions: Drug: Palmitoylethanolamide sold as Levagen +
- A comparator placebo capsule - Maltodextrin and microcrystalline cellulose mix (Placebo Comparator): A comparator capsule taken as a 700mg (2 x 350mg) dosage at onset of migraine and if unresolved at 2 hours post onset a second dose of 700mg (2 x 350mg)
  Interventions: Drug: Placebo comparator - maltodextrin and microcrystalline cellulose mix

INTERVENTIONS:
Drug: Palmitoylethanolamide sold as Levagen + — Investigational product to be taken as a 700mg (2 x 350mg) dosage at onset of migraine. If unresolved at 2 hours post onset of migraine, a second dose of 700mg (2 x 350mg) is to be taken.
  Other Names: Levagen+
  Arms: Palmitoylethanolamide sold as Levagen +
Drug: Placebo comparator - maltodextrin and microcrystalline cellulose mix — Placebo product to be taken as a 700mg (2 x 350mg) dosage at onset of migraine. If unresolved at 2 hours post onset of migraine, a second dose of 700mg (2 x 350mg) is to be taken.
  Arms: A comparator placebo capsule - Maltodextrin and microcrystalline cellulose mix

SUMMARY:
This is a double-blind randomised controlled study to evaluate the effectiveness of orally-dosed Palmitoylethanolamide (PEA) compared to placebo for reducing pain severity and duration of migraines in otherwise healthy participants aged 18 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18
* No recent history (within 2 years) of clinically significant medical conditions including, but not limited to, malignancy (and treatment for malignancy), cardiovascular, neurological, psychiatric, renal, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled*.
* Participant's full agreement and ability to consent to participation in the study
* At least 1 migraine (not headache) episode every 2 months as classified according to the International Classification of Headache Disorders, 3rd edition (ICHD3) for migraines published by the International Headache Society as detailed in section "Classification"
* Access to a computer or smartphone for completing online questionnaires and events.

Exclusion Criteria:

* Use of long-term medication (unless for controlled medical condition as above)
* Pregnant, trying to get pregnant or lactating women^
* Chronic past and/or current alcohol use (greater than 14 alcoholic drinks week)
* Smokers
* Allergic or hypersensitive to any of the ingredients in the active or placebo formula
* Use of preventative migraine medication
* Migraines that have reported:

  * To occur on 15 or more days/month for more than 3 months, which, on at least 8 days/month, has the features of migraine headache.
  * A debilitating attack lasting for more than 72 hours.
  * A seizure

    * A medical condition will be considered uncontrolled if the participant reports ongoing treatment, a change of either medication type or dose in the past 3 months or any change in symptoms within the past 3 months.

      * Any person suspecting they may be pregnant (e.g. missed period, nausea, fatigue) will be directed to attend their GP for a pregnancy test prior to enrolment in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Reduction in migraine pain/severity as assessed by VAS (Visual Analog Scale) for pain Migraine Pain/Severity | Baseline (onset of migraine), 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 2 hours 30 minutes, 3 hours, 3 hour 30 minutes, 4 hours, 5 hours, 6 hours, 7 hours and 8 hours (primary endpoint).
  Change in migraine pain/severity as assessed by VAS (Visual Analog Scale) for pain - Minimum score = 0, Maximum score = 100. Higher scores indicate a higher level of pain/severity.

SECONDARY OUTCOMES:
Migraine Duration | Baseline (onset of migraine), 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 2 hours 30 minutes, 3 hours, 3 hour 30 minutes, 4 hours, 5 hours, 6 hours, 7 hours and 8 hours (primary endpoint).
  Change in migraine duration
Pain relief medication use | Baseline (onset of migraine), 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 2 hours 30 minutes, 3 hours, 3 hour 30 minutes, 4 hours, 5 hours, 6 hours, 7 hours and 8 hours (primary endpoint).
  Change in pain relief medication use

CONTACTS AND LOCATIONS:
Overall Officials: David Briskey, PhD, Principal Investigator — RDC Global Pty Ltd
Locations (1):
- RDC Global Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared